CLINICAL TRIAL: NCT01324011
Title: Family Diabetes Study (Family PALS (PArtners in Lifestyle Support)
Brief Title: Family PALS (PArtners in Lifestyle Support)
Acronym: PALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Carmen Samuel-Hodge, PhD, Research Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-1449; K01DK080079 (NIH)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-based intervention (Experimental): Special intervention (20 weekly group-based sessions) to be compared with a delayed intervention control group.
  Interventions: Behavioral: Adult diabetes family-based weight loss intervention
- Delayed intervention controls (Other): The delayed intervention controls will continue with usual care (if patients with diabetes)and at the end of the experimental period (6 months), they will receive a 6-session weight loss intervention delivered over a 2 month period.
  Interventions: Behavioral: Adult diabetes family-based weight loss intervention

INTERVENTIONS:
Behavioral: Adult diabetes family-based weight loss intervention — Participants assigned to the experimental group will begin the 2o-week weight loss intervention, while delayed intervention controls will wait until the end of this period to begin their program. The weight loss intervention includes 20 weekly group-based sessions facilitated by a registered dietitian. Each group session will last about 120 minutes and include: weight check, group sharing and problem-solving, discussion of a weight control topics (nutrition, physical activity, or behavior change), physical activity and/or taste-testing. Ten sessions will include a brief component, focused on improving family relationships for better diabetes self-care. The study weight loss goal is ≥10 pounds (minimum rate-0.5 lb/week; maximum-2 lbs/week). While the control group waits, they will receive 1 newsletter with study updates and general health or diabetes information. The delayed intervention includes 6 sessions (4 weekly + 2 bi-weekly) following the same format as the experimental group.
  Other Names: intense weight loss intervention; family-based lifestyle intervention

SUMMARY:
NOTE: This study is in the trial-phase of a 5-year study that included a formative research phase (Phase 1 - IRB study # 07-1765 "Family-based Diabetes Self-management Training for African American Adults"). During the first phase, eight focus groups were conducted with 68 participants and a validation study with 215 African American patients with type 2 diabetes. The data gathered in Phase 1 informs the refinement of the intervention in this phase.

Purpose: The overall goal of this research is to evaluate, in a randomized controlled trial, a family-based diabetes self-management intervention for overweight/obese African American adults with type 2 diabetes (the "index participants") and a paired overweight family member (co-participant) who does not have diabetes. The primary outcome is weight change in the index participant.

DETAILED DESCRIPTION:
Type 2 diabetes disproportionately burdens African Americans, and already excessive rates of diabetes are expected to increase even further as rates of obesity rise. While there is evidence that diabetes self-management training is effective in improving metabolic control, and modest weight loss can delay the onset of diabetes, the investigators have limited knowledge of the best approach to self-management training from a family perspective in high risk groups such as African Americans. Family remains a valued dimension of African American life and may be an important behavioral context for interventions to improve disease management and health outcomes. Nonetheless, there are no trials of family-based interventions to improve diabetes self-care and achieve weight loss that have involved adult families.

Participants: A total of 80 pairs (index participant + family member) or 160 adults will participate in this trial where a 20-session behavioral weight loss intervention will be tested. Participants include overweight or obese African Americans with type 2 diabetes and a paired co-participant identified as an overweight or obese adult family member without type 2 diabetes. Family members may self-describe as non-African Americans.

Procedures (methods): Study participants will be enrolled in a randomized controlled trial using a 2:1 random allocation to the special intervention (a 20-session family-based behavioral weight loss intervention) or a usual care group (controls). Following the trial, participants in the usual care group will receive a 6-session weight management intervention (over a 2-month period) based on the 20-session special intervention.

ELIGIBILITY:
Person with diabetes.

Inclusion Criteria:

* self-described African American 21-75 years of age;
* self-reported diagnosis of type 2 diabetes;
* A1c value ≤ 11%;
* currently under the care of a physician or other health care provider;
* able to participate in moderate level physical activity;
* willing to lose 5% or more of initial body weight and follow recommendations for healthy dietary and physical activity patterns;
* access to a phone and willing to complete a telephone-administered survey;
* English speaking.

Exclusion Criteria:

* any medical contraindication to weight loss;
* cardiovascular event within the past 6 months;
* evidence of active cancer diagnosis;
* pregnant or lactating;
* self-reported history of renal disease other than kidney stones;
* any history of gastric bypass surgery or scheduled surgery for this purpose;
* weight loss of >20 lbs in the last 3 months;
* current use of medications for weight loss, treatment of psychosis or manic-depressive illness.

Family Members: Inclusion criteria (NOTE: 'Family' for this study is defined as 'a group of intimates living together or in close proximity with strong emotional bonds (identification, attachment, loyalty, reciprocity, solidarity), and with strong, ongoing personal ties. Family members can only participate if paired with an African American study participant.):

* 21 -75 years of age;
* living with or married (for at least 1 year) to an African American adult diagnosed with diabetes;
* self-described as a blood relative of an African American with diabetes with whom there is regular, ongoing contact;
* overweight/obesity defined as a BMI between 25 to 47, inclusive;
* English-speaking;
* able to participate in moderate level physical activity;
* willing to lose 5% or more of initial body weight and follow recommendations for healthy dietary and physical activity patterns;
* access to a phone and willing to complete a telephone-administered survey.

Exclusion Criteria:

* self-reported diagnosis of type 2 diabetes (the A1c test used in this study cannot be used for diagnostic purposes; additionally, the initial therapy of most newly diagnosed patients with type 2 diabetes includes lifestyle changes and weight loss);
* any medical contraindication to weight loss;
* cardiovascular event within the past 6 months;
* evidence of active cancer diagnosis;
* pregnant or lactating;
* self-reported history of renal disease other than kidney stones;
* any history of gastric bypass surgery or scheduled surgery for this purpose;
* weight loss of > 20 lbs in the last 3 months;
* current use of medications for weight loss, treatment of psychosis or manic-depressive illness.

Family members do not themselves have to be self-described African Americans.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 6 months
  Change in weight from start to end of the 20-weekly group-based intervention. NOTE: Weekly sessions are not held during weeks where holidays occur on a scheduled session date (such that the duration of the intervention may be more than 20 weeks).

SECONDARY OUTCOMES:
Effect on Hemoglobin A1c | 6 months (post-intervention)
  A1c change from enrollment to post-intervention.
Lifestyle behaviors | 6 months
  Diet and physical activity behavior changes (from enrollment or baseline to post-intervention)
Blood pressure change | 6 months
  Change in systolic and diastolic blood pressure from baseline (enrollment) to post-intervention
Change in psychosocial factors | 6 months
  Changes in measures of family functioning, social support and social relationships, self-efficacy, perceived barriers to diabetes self-care, and quality of life; comparing baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen D. Samuel-Hodge, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Health Promotion and Disease Prevention (HPDP), Chapel Hill, North Carolina, United States